CLINICAL TRIAL: NCT04890067
Title: Multicenter Observational Study on the Treatment of Patients With Localized Osteosarcoma
Brief Title: Observational Study in Localized Osteosarcoma
Acronym: ISG Os2Oss
Status: Recruiting | Type: Observational
Sponsor: Italian Sarcoma Group (Network)
Collaborators: Associazione Italiana Ematologia Oncologia Pediatrica (Other)
Responsible Party: Sponsor
Other Study IDs: AIEOP/ISGOS2 Oss
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Localized Osteosarcoma
Keywords: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Localized Osteosarcoma: This cohort include patients affected by localized Osteosarcoma, referred to participating Institutions.
  Interventions: Other: Treatment of Osteosarcoma according the AIEOP/ISG OS 2021 recommendations (includes drugs, surgery, radiotherapy or any other received treatments)

INTERVENTIONS:
Other: Treatment of Osteosarcoma according the AIEOP/ISG OS 2021 recommendations (includes drugs, surgery, radiotherapy or any other received treatments) — This observational study collects all the treatments received by the patients according according the AIEOP/ISG OS 2021 and therefore includes drug/biological/surgical/ radiotherapy and any other applicable treatments

SUMMARY:
Observational prospective trial aimed to collect the collect demographic, clinical, surgical, pathological and molecular characteristics and treatment from patients affected by localized OsteoSarcoma (OS) treated according the AIEOP/Italian Sarcoma Group (ISG) OS 2021

DETAILED DESCRIPTION:
Osteosarcoma is the most frequent primary malignant bone tumor in children and adolescents and is considered a rare disease.

The overall incidence of OS is 0.2-3 / 100,000 inhabitants per year with a bimodal distribution by age, with a first peak in adolescence.

Currently, the treatment strategy for localized OS includes courses of neo-adjuvant chemotherapy based on 3 agents: Adriamycin (ADM), cisplatin (CDP) and high dose methotrexate (HDMTX) followed by surgical removal of the primary tumor and subsequent adjuvant chemotherapy treatment.

The MAP (Methotrexate, Adriamycin, cisPlatin) regimen, with or without ifosfamide (IFO) and etoposide (ETO), is considered the "gold standard" for the treatment of localized osteosarcoma.

Given the rarity of the disease, it is considered appropriate to collect information prospectively on the diagnosis, chemotherapy and surgical treatment and outcomes on patients treated by the network of AIEOP and ISG Centers according to the recommendations on the treatment of localized OS AIEOP/ISG OS 2021.

This study will be active up to the next interventional prospective protocol aimed at the therapy of high-grade, non-metastatic OS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high grade OS of the extremities
* Age at diagnosis ≤ 40 years at the time of diagnosis
* Localized disease (skip metastases are allowed)
* Adequate organ function according the AIEOP/ISG OS 2021 recommendation
* Patients or parents oe guardians of minors who have given their written informed consent to participate in the study

Exclusion Criteria:

* Presence of metastases
* Diagnosis of periosteal OS, of parosteal OS or secondary OS
* Any medical condition which can not allowed the use of the treatments recommended by AIEOP/ISG OS 2021

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with localized high grade ostesarcoma of the extremities
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
5 years Event Free Survival (EFS) | 5 years
  Onset of any event (an event is the defined as disease recurrence, death for disease or any other cause)

SECONDARY OUTCOMES:
Overall Survival (OS) | at 5 years
  Time elapsed for the diagnosis to the death for any cause
Adverse events related to the treatments | Every 3 weeks (Week 3, week 6, week 9, week 12, ...) up to 36 months
  Number of Participants with Treatment-Related Adverse Events as Assessed by Common Terminology Criteria for Adverse Events version 5.0

CONTACTS AND LOCATIONS:
Locations (16):
- Italy (16):
  - Centro di Riferimento Oncologico - Unit of Medical Oncology, Aviano, Pordenone
  - Sandra Aliberti, Candiolo, Torino
  - IRCCS materno infantile Burlo Garofolo, Trieste, T
  - Azienda Ospedaliero Universitaria Consorziale Policlinico - Bari, Bari
  - IRCCS Istituto ortopedico Rizzoli, Bologna
  - A.O. Universitaria Policlinico S. Orsola Malpighi di Bologna, Bologna
  - AUO Policnico G. Rodolico San Marco, Catania
  - A.O. Universitaria Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS INT Milano SC Pediatria Oncologica, Milan
  - FONDAZIONE IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera di Padova UOC Oncoematologia Pediatrica, Padua
  - ARNAS P. O. "Civico e Benfratelli", Palermo
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Istituti Fisioterapici Ospitalieri di Roma, Roma
  - Ospedale Pediatrico Bambin Gesu', Roma

IPD SHARING:
Plan to Share IPD: No
No plan sharing

REFERENCES:
- [Background] Mirabello L, Troisi RJ, Savage SA. Osteosarcoma incidence and survival rates from 1973 to 2004: data from the Surveillance, Epidemiology, and End Results Program. Cancer. 2009 Apr 1;115(7):1531-43. doi: 10.1002/cncr.24121. PMID 19197972
- [Background] Marina N, Gebhardt M, Teot L, Gorlick R. Biology and therapeutic advances for pediatric osteosarcoma. Oncologist. 2004;9(4):422-41. doi: 10.1634/theoncologist.9-4-422. PMID 15266096
- [Background] Casali PG, Bielack S, Abecassis N, Aro HT, Bauer S, Biagini R, Bonvalot S, Boukovinas I, Bovee JVMG, Brennan B, Brodowicz T, Broto JM, Brugieres L, Buonadonna A, De Alava E, Dei Tos AP, Del Muro XG, Dileo P, Dhooge C, Eriksson M, Fagioli F, Fedenko A, Ferraresi V, Ferrari A, Ferrari S, Frezza AM, Gaspar N, Gasperoni S, Gelderblom H, Gil T, Grignani G, Gronchi A, Haas RL, Hassan B, Hecker-Nolting S, Hohenberger P, Issels R, Joensuu H, Jones RL, Judson I, Jutte P, Kaal S, Kager L, Kasper B, Kopeckova K, Krakorova DA, Ladenstein R, Le Cesne A, Lugowska I, Merimsky O, Montemurro M, Morland B, Pantaleo MA, Piana R, Picci P, Piperno-Neumann S, Pousa AL, Reichardt P, Robinson MH, Rutkowski P, Safwat AA, Schoffski P, Sleijfer S, Stacchiotti S, Strauss SJ, Sundby Hall K, Unk M, Van Coevorden F, van der Graaf WTA, Whelan J, Wardelmann E, Zaikova O, Blay JY; ESMO Guidelines Committee, PaedCan and ERN EURACAN. Bone sarcomas: ESMO-PaedCan-EURACAN Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv79-iv95. doi: 10.1093/annonc/mdy310. No abstract available. PMID 30285218
- [Background] Ottaviani G, Jaffe N. The epidemiology of osteosarcoma. Cancer Treat Res. 2009;152:3-13. doi: 10.1007/978-1-4419-0284-9_1. PMID 20213383
- [Background] Gatta G, Botta L, Rossi S, Aareleid T, Bielska-Lasota M, Clavel J, Dimitrova N, Jakab Z, Kaatsch P, Lacour B, Mallone S, Marcos-Gragera R, Minicozzi P, Sanchez-Perez MJ, Sant M, Santaquilani M, Stiller C, Tavilla A, Trama A, Visser O, Peris-Bonet R; EUROCARE Working Group. Childhood cancer survival in Europe 1999-2007: results of EUROCARE-5--a population-based study. Lancet Oncol. 2014 Jan;15(1):35-47. doi: 10.1016/S1470-2045(13)70548-5. Epub 2013 Dec 5. PMID 24314616
- [Background] Mirabello L, Troisi RJ, Savage SA. International osteosarcoma incidence patterns in children and adolescents, middle ages and elderly persons. Int J Cancer. 2009 Jul 1;125(1):229-34. doi: 10.1002/ijc.24320. PMID 19330840
- [Background] Geller DS, Gorlick R. Osteosarcoma: a review of diagnosis, management, and treatment strategies. Clin Adv Hematol Oncol. 2010 Oct;8(10):705-18. PMID 21317869
- [Background] Bielack SS, Kempf-Bielack B, Delling G, Exner GU, Flege S, Helmke K, Kotz R, Salzer-Kuntschik M, Werner M, Winkelmann W, Zoubek A, Jurgens H, Winkler K. Prognostic factors in high-grade osteosarcoma of the extremities or trunk: an analysis of 1,702 patients treated on neoadjuvant cooperative osteosarcoma study group protocols. J Clin Oncol. 2002 Feb 1;20(3):776-90. doi: 10.1200/JCO.2002.20.3.776. PMID 11821461
- [Background] Luetke A, Meyers PA, Lewis I, Juergens H. Osteosarcoma treatment - where do we stand? A state of the art review. Cancer Treat Rev. 2014 May;40(4):523-32. doi: 10.1016/j.ctrv.2013.11.006. Epub 2013 Nov 27. PMID 24345772
- [Background] Ferrari S, Ruggieri P, Cefalo G, Tamburini A, Capanna R, Fagioli F, Comandone A, Bertulli R, Bisogno G, Palmerini E, Alberghini M, Parafioriti A, Linari A, Picci P, Bacci G. Neoadjuvant chemotherapy with methotrexate, cisplatin, and doxorubicin with or without ifosfamide in nonmetastatic osteosarcoma of the extremity: an Italian sarcoma group trial ISG/OS-1. J Clin Oncol. 2012 Jun 10;30(17):2112-8. doi: 10.1200/JCO.2011.38.4420. Epub 2012 May 7. PMID 22564997
- [Background] Ferrari S, Meazza C, Palmerini E, Tamburini A, Fagioli F, Cozza R, Ferraresi V, Bisogno G, Mascarin M, Cefalo G, Manfrini M, Capanna R, Biagini R, Donati D, Picci P. Nonmetastatic osteosarcoma of the extremity. Neoadjuvant chemotherapy with methotrexate, cisplatin, doxorubicin and ifosfamide. An Italian Sarcoma Group study (ISG/OS-Oss). Tumori. 2014 Nov-Dec;100(6):612-9. doi: 10.1700/1778.19262. PMID 25688494
- [Background] Meyers PA, Schwartz CL, Krailo MD, Healey JH, Bernstein ML, Betcher D, Ferguson WS, Gebhardt MC, Goorin AM, Harris M, Kleinerman E, Link MP, Nadel H, Nieder M, Siegal GP, Weiner MA, Wells RJ, Womer RB, Grier HE; Children's Oncology Group. Osteosarcoma: the addition of muramyl tripeptide to chemotherapy improves overall survival--a report from the Children's Oncology Group. J Clin Oncol. 2008 Feb 1;26(4):633-8. doi: 10.1200/JCO.2008.14.0095. PMID 18235123
- [Background] Bacci G, Picci P, Ferrari S, Sangiorgi L, Zanone A, Brach del Prever A. Primary chemotherapy and delayed surgery for non-metastatic telangiectatic osteosarcoma of the extremities. Results in 28 patients. Eur J Cancer. 1994;30A(5):620-6. doi: 10.1016/0959-8049(94)90532-0. PMID 8080676
- [Background] Bacci G, Ferrari S, Mercuri M, Longhi A, Capanna R, Tienghi A, Brach del Prever A, Comandone A, Cesari M, Bernini G, Picci P. Neoadjuvant chemotherapy for extremity osteosarcoma--preliminary results of the Rizzoli's 4th study. Acta Oncol. 1998;37(1):41-8. doi: 10.1080/028418698423168. PMID 9572653
- [Background] Ferrari S, Smeland S, Mercuri M, Bertoni F, Longhi A, Ruggieri P, Alvegard TA, Picci P, Capanna R, Bernini G, Muller C, Tienghi A, Wiebe T, Comandone A, Bohling T, Del Prever AB, Brosjo O, Bacci G, Saeter G; Italian and Scandinavian Sarcoma Groups. Neoadjuvant chemotherapy with high-dose Ifosfamide, high-dose methotrexate, cisplatin, and doxorubicin for patients with localized osteosarcoma of the extremity: a joint study by the Italian and Scandinavian Sarcoma Groups. J Clin Oncol. 2005 Dec 1;23(34):8845-52. doi: 10.1200/JCO.2004.00.5785. Epub 2005 Oct 24. PMID 16246977
- [Background] Smeland S, Muller C, Alvegard TA, Wiklund T, Wiebe T, Bjork O, Stenwig AE, Willen H, Holmstrom T, Folleras G, Brosjo O, Kivioja A, Jonsson K, Monge O, Saeter G. Scandinavian Sarcoma Group Osteosarcoma Study SSG VIII: prognostic factors for outcome and the role of replacement salvage chemotherapy for poor histological responders. Eur J Cancer. 2003 Mar;39(4):488-94. doi: 10.1016/s0959-8049(02)00747-5. PMID 12751380
- [Background] Le Deley MC, Guinebretiere JM, Gentet JC, Pacquement H, Pichon F, Marec-Berard P, Entz-Werle N, Schmitt C, Brugieres L, Vanel D, Dupouy N, Tabone MD, Kalifa C; Societe Francaise d'Oncologie Pediatrique (SFOP). SFOP OS94: a randomised trial comparing preoperative high-dose methotrexate plus doxorubicin to high-dose methotrexate plus etoposide and ifosfamide in osteosarcoma patients. Eur J Cancer. 2007 Mar;43(4):752-61. doi: 10.1016/j.ejca.2006.10.023. Epub 2007 Jan 30. PMID 17267204
- [Background] Piperno-Neumann S, Le Deley MC, Redini F, Pacquement H, Marec-Berard P, Petit P, Brisse H, Lervat C, Gentet JC, Entz-Werle N, Italiano A, Corradini N, Bompas E, Penel N, Tabone MD, Gomez-Brouchet A, Guinebretiere JM, Mascard E, Gouin F, Chevance A, Bonnet N, Blay JY, Brugieres L; Sarcoma Group of UNICANCER; French Society of Pediatric Oncology (SFCE); French Sarcoma Group (GSF-GETO). Zoledronate in combination with chemotherapy and surgery to treat osteosarcoma (OS2006): a randomised, multicentre, open-label, phase 3 trial. Lancet Oncol. 2016 Aug;17(8):1070-1080. doi: 10.1016/S1470-2045(16)30096-1. Epub 2016 Jun 17. PMID 27324280
- [Background] Smeland S, Bielack SS, Whelan J, Bernstein M, Hogendoorn P, Krailo MD, Gorlick R, Janeway KA, Ingleby FC, Anninga J, Antal I, Arndt C, Brown KLB, Butterfass-Bahloul T, Calaminus G, Capra M, Dhooge C, Eriksson M, Flanagan AM, Friedel G, Gebhardt MC, Gelderblom H, Goldsby R, Grier HE, Grimer R, Hawkins DS, Hecker-Nolting S, Sundby Hall K, Isakoff MS, Jovic G, Kuhne T, Kager L, von Kalle T, Kabickova E, Lang S, Lau CC, Leavey PJ, Lessnick SL, Mascarenhas L, Mayer-Steinacker R, Meyers PA, Nagarajan R, Randall RL, Reichardt P, Renard M, Rechnitzer C, Schwartz CL, Strauss S, Teot L, Timmermann B, Sydes MR, Marina N. Survival and prognosis with osteosarcoma: outcomes in more than 2000 patients in the EURAMOS-1 (European and American Osteosarcoma Study) cohort. Eur J Cancer. 2019 Mar;109:36-50. doi: 10.1016/j.ejca.2018.11.027. Epub 2019 Jan 25. PMID 30685685
- [Background] Rosen G, Caparros B, Huvos AG, Kosloff C, Nirenberg A, Cacavio A, Marcove RC, Lane JM, Mehta B, Urban C. Preoperative chemotherapy for osteogenic sarcoma: selection of postoperative adjuvant chemotherapy based on the response of the primary tumor to preoperative chemotherapy. Cancer. 1982 Mar 15;49(6):1221-30. doi: 10.1002/1097-0142(19820315)49:63.0.co;2-e. PMID 6174200
- [Background] Ferrari S, Bacci G, Picci P, Mercuri M, Briccoli A, Pinto D, Gasbarrini A, Tienghi A, Brach del Prever A. Long-term follow-up and post-relapse survival in patients with non-metastatic osteosarcoma of the extremity treated with neoadjuvant chemotherapy. Ann Oncol. 1997 Aug;8(8):765-71. doi: 10.1023/a:1008221713505. PMID 9332684
- [Background] Bishop MW, Chang YC, Krailo MD, Meyers PA, Provisor AJ, Schwartz CL, Marina NM, Teot LA, Gebhardt MC, Gorlick R, Janeway KA, Chou AJ. Assessing the Prognostic Significance of Histologic Response in Osteosarcoma: A Comparison of Outcomes on CCG-782 and INT0133-A Report From the Children's Oncology Group Bone Tumor Committee. Pediatr Blood Cancer. 2016 Oct;63(10):1737-43. doi: 10.1002/pbc.26034. Epub 2016 Apr 29. PMID 27128693
- [Background] Harrison DJ, Geller DS, Gill JD, Lewis VO, Gorlick R. Current and future therapeutic approaches for osteosarcoma. Expert Rev Anticancer Ther. 2018 Jan;18(1):39-50. doi: 10.1080/14737140.2018.1413939. Epub 2017 Dec 14. PMID 29210294
- [Background] Nardin A, Lefebvre ML, Labroquere K, Faure O, Abastado JP. Liposomal muramyl tripeptide phosphatidylethanolamine: Targeting and activating macrophages for adjuvant treatment of osteosarcoma. Curr Cancer Drug Targets. 2006 Mar;6(2):123-33. doi: 10.2174/156800906776056473. PMID 16529542
- [Background] Kleinerman ES, Erickson KL, Schroit AJ, Fogler WE, Fidler IJ. Activation of tumoricidal properties in human blood monocytes by liposomes containing lipophilic muramyl tripeptide. Cancer Res. 1983 May;43(5):2010-4. PMID 6831430
- [Background] Anderson P. Liposomal muramyl tripeptide phosphatidyl ethanolamine: ifosfamide-containing chemotherapy in osteosarcoma. Future Oncol. 2006 Jun;2(3):333-43. doi: 10.2217/14796694.2.3.333. PMID 16787112
- [Background] Isakoff MS, Bielack SS, Meltzer P, Gorlick R. Osteosarcoma: Current Treatment and a Collaborative Pathway to Success. J Clin Oncol. 2015 Sep 20;33(27):3029-35. doi: 10.1200/JCO.2014.59.4895. Epub 2015 Aug 24. PMID 26304877
- [Background] Meyers PA, Schwartz CL, Krailo M, Kleinerman ES, Betcher D, Bernstein ML, Conrad E, Ferguson W, Gebhardt M, Goorin AM, Harris MB, Healey J, Huvos A, Link M, Montebello J, Nadel H, Nieder M, Sato J, Siegal G, Weiner M, Wells R, Wold L, Womer R, Grier H. Osteosarcoma: a randomized, prospective trial of the addition of ifosfamide and/or muramyl tripeptide to cisplatin, doxorubicin, and high-dose methotrexate. J Clin Oncol. 2005 Mar 20;23(9):2004-11. doi: 10.1200/JCO.2005.06.031. PMID 15774791
- [Background] Ando K, Mori K, Corradini N, Redini F, Heymann D. Mifamurtide for the treatment of nonmetastatic osteosarcoma. Expert Opin Pharmacother. 2011 Feb;12(2):285-92. doi: 10.1517/14656566.2011.543129. PMID 21226638
- [Background] Marina N, Bielack S, Whelan J, Smeland S, Krailo M, Sydes MR, Butterfass-Bahloul T, Calaminus G, Bernstein M. International collaboration is feasible in trials for rare conditions: the EURAMOS experience. Cancer Treat Res. 2009;152:339-53. doi: 10.1007/978-1-4419-0284-9_18. PMID 20213400
- [Background] Bishop MW, Janeway KA, Gorlick R. Future directions in the treatment of osteosarcoma. Curr Opin Pediatr. 2016 Feb;28(1):26-33. doi: 10.1097/MOP.0000000000000298. PMID 26626558
- [Background] Marina NM, Smeland S, Bielack SS, Bernstein M, Jovic G, Krailo MD, Hook JM, Arndt C, van den Berg H, Brennan B, Brichard B, Brown KLB, Butterfass-Bahloul T, Calaminus G, Daldrup-Link HE, Eriksson M, Gebhardt MC, Gelderblom H, Gerss J, Goldsby R, Goorin A, Gorlick R, Grier HE, Hale JP, Hall KS, Hardes J, Hawkins DS, Helmke K, Hogendoorn PCW, Isakoff MS, Janeway KA, Jurgens H, Kager L, Kuhne T, Lau CC, Leavey PJ, Lessnick SL, Mascarenhas L, Meyers PA, Mottl H, Nathrath M, Papai Z, Randall RL, Reichardt P, Renard M, Safwat AA, Schwartz CL, Stevens MCG, Strauss SJ, Teot L, Werner M, Sydes MR, Whelan JS. Comparison of MAPIE versus MAP in patients with a poor response to preoperative chemotherapy for newly diagnosed high-grade osteosarcoma (EURAMOS-1): an open-label, international, randomised controlled trial. Lancet Oncol. 2016 Oct;17(10):1396-1408. doi: 10.1016/S1470-2045(16)30214-5. Epub 2016 Aug 25. PMID 27569442
- [Background] Serra M, Scotlandi K, Reverter-Branchat G, Ferrari S, Manara MC, Benini S, Incaprera M, Bertoni F, Mercuri M, Briccoli A, Bacci G, Picci P. Value of P-glycoprotein and clinicopathologic factors as the basis for new treatment strategies in high-grade osteosarcoma of the extremities. J Clin Oncol. 2003 Feb 1;21(3):536-42. doi: 10.1200/JCO.2003.03.144. PMID 12560446
- [Background] Serra M, Pasello M, Manara MC, Scotlandi K, Ferrari S, Bertoni F, Mercuri M, Alvegard TA, Picci P, Bacci G, Smeland S. May P-glycoprotein status be used to stratify high-grade osteosarcoma patients? Results from the Italian/Scandinavian Sarcoma Group 1 treatment protocol. Int J Oncol. 2006 Dec;29(6):1459-68. PMID 17088985